CLINICAL TRIAL: NCT02692716
Title: A Trial Investigating the Cardiovascular Safety of Oral Semaglutide in Subjects With Type 2 Diabetes
Acronym: PIONEER 6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9924-4221; 2015-003563-10 (EudraCT Number); U1111-1173-0750 (Other: WHO); NL56580.091.16 (Other: CCMO)
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral semaglutide (Experimental)
  Interventions: Drug: semaglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: semaglutide — For oral use once daily.
  Arms: Oral semaglutide
Drug: placebo — For oral use once daily.
  Arms: Placebo

SUMMARY:
This trial is conducted globally. The aim of the trial is to investigate the cardiovascular safety of oral semaglutide in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female diagnosed with type 2 diabetes
* Age at least 50 years at screening and presence of cardiovascular disease, or age at least 60 years at screening and presence of at least one cardiovascular risk factor

Exclusion Criteria:

* Current or previous (within 90 days prior to screening) treatment with any GLP-1 (glucagon-like peptide-1) receptor agonist, DPP-4 (dipeptidyl peptidase-4) inhibitor or pramlintide
* Family or personal history of multiple endocrine neoplasia type 2 (MEN 2) or medullary thyroid carcinoma (MTC)
* History of pancreatitis (acute or chronic)
* History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery)
* Subjects presently classified as being in New York Heart Association (NYHA) Class IV heart failure
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening
* Any of the following: myocardial infarction, stroke or hospitalisation for unstable angina or transient ischaemic attack within the past 60 days prior to screening
* Chronic or intermittent hemodialysis or peritoneal dialysis or severe renal impairment (corresponding to eGFR (glomerular filtration rate, estimated) below 30 mL/min/1.73 m^2)
* History or presence of malignant neoplasms within the last 5 years (except basal and squamous cell skin cancer and carcinoma in situ)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3183 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (191):
- United States (61):
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, Searcy, Arkansas
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Huntington Beach, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, La Mesa, California
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, Monterey, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, San Ramon, California
  - Novo Nordisk Investigational Site, Ventura, California
  - Novo Nordisk Investigational Site, Boca Raton, Florida
  - Novo Nordisk Investigational Site, New Port Richey, Florida
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Savannah, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Michigan City, Indiana
  - Novo Nordisk Investigational Site, Muncie, Indiana
  - Novo Nordisk Investigational Site, Council Bluffs, Iowa
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Monroe, Louisiana
  - Novo Nordisk Investigational Site, Slidell, Louisiana
  - Novo Nordisk Investigational Site, Canton, Michigan
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, North Massapequa, New York
  - Novo Nordisk Investigational Site, Westfield, New York
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Fargo, North Dakota
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Maumee, Ohio
  - Novo Nordisk Investigational Site, Beaver, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Anderson, South Carolina
  - Novo Nordisk Investigational Site, Moncks Corner, South Carolina
  - Novo Nordisk Investigational Site, Myrtle Beach, South Carolina
  - Novo Nordisk Investigational Site, Spartanburg, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Knoxville, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Hurst, Texas
  - Novo Nordisk Investigational Site, Midland, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Waco, Texas
  - Novo Nordisk Investigational Site, South Burlington, Vermont
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Winchester, Virginia
- Algeria (4):
  - Novo Nordisk Investigational Site, Annaba
  - Novo Nordisk Investigational Site, Oran
  - Novo Nordisk Investigational Site, Sétif
  - Novo Nordisk Investigational Site, Tizi Ouzou
- Argentina (4):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, CABA
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Lanús Este
- Brazil (4):
  - Novo Nordisk Investigational Site, Curitiba, Paraná
  - Novo Nordisk Investigational Site, Mogi das Cruzes, São Paulo
  - Novo Nordisk Investigational Site, São José dos Campos, São Paulo
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
- Canada (6):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Brampton, Ontario
  - Novo Nordisk Investigational Site, Concord, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Montreal, Quebec
- Denmark (5):
  - Novo Nordisk Investigational Site, Aarhus N
  - Novo Nordisk Investigational Site, Esbjerg
  - Novo Nordisk Investigational Site, Hellerup
  - Novo Nordisk Investigational Site, Hvidovre
  - Novo Nordisk Investigational Site, Odense
- Germany (12):
  - Novo Nordisk Investigational Site, Bochum
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Elsterwerda
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Oldenburg
  - Novo Nordisk Investigational Site, Oldenburg I. Holst
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
- India (15):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Hyderbad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Kochi, Kerala
  - Novo Nordisk Investigational Site, Kozhikode, Kerala
  - Novo Nordisk Investigational Site, Thiruvananthapuram, Kerala
  - Novo Nordisk Investigational Site, Goa, Maharashtra
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Ludhiana, Punjab
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, New Delhi
  - Novo Nordisk Investigational Site, Pune
- Israel (7):
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Holon
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Nahariya
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Rishon LeZiyyon
  - Novo Nordisk Investigational Site, Tel Aviv
- Italy (6):
  - Novo Nordisk Investigational Site, Bergamo
  - Novo Nordisk Investigational Site, Catanzaro
  - Novo Nordisk Investigational Site, Chieti
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Palermo
  - Novo Nordisk Investigational Site, Roma
- Malaysia (9):
  - Novo Nordisk Investigational Site, Ipoh, Perak
  - Novo Nordisk Investigational Site, Kota Bharu
  - Novo Nordisk Investigational Site, Kota Bharu, Kelantan
  - Novo Nordisk Investigational Site, Kota Samarahan
  - Novo Nordisk Investigational Site, Kuala Lumpur
  - Novo Nordisk Investigational Site, Kuching
  - Novo Nordisk Investigational Site, Malacca
  - Novo Nordisk Investigational Site, Putrajaya
  - Novo Nordisk Investigational Site, Seremban
- Mexico (4):
  - Novo Nordisk Investigational Site, Guadalajara, Jalisco
  - Novo Nordisk Investigational Site, Monterrey, Nuevo León
  - Novo Nordisk Investigational Site, Mérida, Yucatán
  - Novo Nordisk Investigational Site, San Luis Potosí City
- Netherlands (5):
  - Novo Nordisk Investigational Site, Almere Stad
  - Novo Nordisk Investigational Site, Amsterdam
  - Novo Nordisk Investigational Site, Eindhoven
  - Novo Nordisk Investigational Site, Hoogeveen
  - Novo Nordisk Investigational Site, Nijmegen
- Poland (4):
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Warsaw
- Romania (4):
  - Novo Nordisk Investigational Site, Oradea, Bihor County
  - Novo Nordisk Investigational Site, Târgu Mureş, Mureș County
  - Novo Nordisk Investigational Site, Bucharest
  - Novo Nordisk Investigational Site, Galati
- South Africa (7):
  - Novo Nordisk Investigational Site, Bloemfontein, Free State
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Lenasia, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Middleburg, Mpumalanga
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
- Spain (9):
  - Novo Nordisk Investigational Site, Alcalá de Henares
  - Novo Nordisk Investigational Site, Badalona
  - Novo Nordisk Investigational Site, Fuenlabrada - Madrid
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Pontevedra
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia
- Taiwan (4):
  - Novo Nordisk Investigational Site, Kaohsiung City
  - Novo Nordisk Investigational Site, Taichung
  - Novo Nordisk Investigational Site, Tainan
  - Novo Nordisk Investigational Site, Taipei
- Thailand (4):
  - Novo Nordisk Investigational Site, Bangkok
  - Novo Nordisk Investigational Site, Chiang Mai
  - Novo Nordisk Investigational Site, Klong Luang, Pathumthani
  - Novo Nordisk Investigational Site, Nakhon Ratchasima
- Turkey (Türkiye) (8):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Aydin
  - Novo Nordisk Investigational Site, Denizli
  - Novo Nordisk Investigational Site, Gaziantep
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Izmir
  - Novo Nordisk Investigational Site, Rize
- United Kingdom (9):
  - Novo Nordisk Investigational Site, Aberdeen
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Exeter
  - Novo Nordisk Investigational Site, Guildford
  - Novo Nordisk Investigational Site, Norfolk
  - Novo Nordisk Investigational Site, Swansea
  - Novo Nordisk Investigational Site, Watford

REFERENCES:
- [Result] Cefalu WT, Kaul S, Gerstein HC, Holman RR, Zinman B, Skyler JS, Green JB, Buse JB, Inzucchi SE, Leiter LA, Raz I, Rosenstock J, Riddle MC. Cardiovascular Outcomes Trials in Type 2 Diabetes: Where Do We Go From Here? Reflections From a Diabetes Care Editors' Expert Forum. Diabetes Care. 2018 Jan;41(1):14-31. doi: 10.2337/dci17-0057. PMID 29263194
- [Result] Bain SC, Mosenzon O, Arechavaleta R, Bogdanski P, Comlekci A, Consoli A, Deerochanawong C, Dungan K, Faingold MC, Farkouh ME, Franco DR, Gram J, Guja C, Joshi P, Malek R, Merino-Torres JF, Nauck MA, Pedersen SD, Sheu WH, Silver RJ, Tack CJ, Tandon N, Jeppesen OK, Strange M, Thomsen M, Husain M. Cardiovascular safety of oral semaglutide in patients with type 2 diabetes: Rationale, design and patient baseline characteristics for the PIONEER 6 trial. Diabetes Obes Metab. 2019 Mar;21(3):499-508. doi: 10.1111/dom.13553. Epub 2018 Nov 11. PMID 30284349
- [Result] Husain M, Birkenfeld AL, Donsmark M, Dungan K, Eliaschewitz FG, Franco DR, Jeppesen OK, Lingvay I, Mosenzon O, Pedersen SD, Tack CJ, Thomsen M, Vilsboll T, Warren ML, Bain SC; PIONEER 6 Investigators. Oral Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. N Engl J Med. 2019 Aug 29;381(9):841-851. doi: 10.1056/NEJMoa1901118. Epub 2019 Jun 11. PMID 31185157
- [Result] Evans LM, Mellbin L, Johansen P, Lawson J, Paine A, Sandberg A. A population-adjusted indirect comparison of cardiovascular benefits of once-weekly subcutaneous semaglutide and dulaglutide in the treatment of patients with type 2 diabetes, with or without established cardiovascular disease. Endocrinol Diabetes Metab. 2021 May 15;4(3):e00259. doi: 10.1002/edm2.259. eCollection 2021 Jul. PMID 34277983
- [Result] Husain M, Consoli A, De Remigis A, Pettersson Meyer AS, Rasmussen S, Bain S. Semaglutide reduces cardiovascular events regardless of metformin use: a post hoc subgroup analysis of SUSTAIN 6 and PIONEER 6. Cardiovasc Diabetol. 2022 Apr 28;21(1):64. doi: 10.1186/s12933-022-01489-6. PMID 35484580
- [Result] Aroda VR, Bauer R, Christiansen E, Haluzik M, Kallenbach K, Montanya E, Rosenstock J, Meier JJ. Efficacy and safety of oral semaglutide by subgroups of patient characteristics in the PIONEER phase 3 programme. Diabetes Obes Metab. 2022 Jul;24(7):1338-1350. doi: 10.1111/dom.14710. Epub 2022 May 9. PMID 35373893
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Bain SC, Belmar N, Hoff ST, Husain M, Rasmussen S, Vilsboll T, Petrie MC. Cardiovascular, Metabolic, and Safety Outcomes with Semaglutide by Baseline Age: Post Hoc Analysis of SUSTAIN 6 and PIONEER 6. Diabetes Ther. 2025 Jan;16(1):15-28. doi: 10.1007/s13300-024-01659-7. Epub 2024 Nov 9. PMID 39520501
- [Derived] Rossing P, Bain SC, Bosch-Traberg H, Sokareva E, Heerspink HJL, Rasmussen S, Mellbin LG. Effect of semaglutide on major adverse cardiovascular events by baseline kidney parameters in participants with type 2 diabetes and at high risk of cardiovascular disease: SUSTAIN 6 and PIONEER 6 post hoc pooled analysis. Cardiovasc Diabetol. 2023 Aug 24;22(1):220. doi: 10.1186/s12933-023-01949-7. PMID 37620807
- [Derived] Strain WD, Frenkel O, James MA, Leiter LA, Rasmussen S, Rothwell PM, Sejersten Ripa M, Truelsen TC, Husain M. Effects of Semaglutide on Stroke Subtypes in Type 2 Diabetes: Post Hoc Analysis of the Randomized SUSTAIN 6 and PIONEER 6. Stroke. 2022 Sep;53(9):2749-2757. doi: 10.1161/STROKEAHA.121.037775. Epub 2022 May 18. PMID 35582947
- [Derived] Verma S, Fainberg U, Husain M, Rasmussen S, Ryden L, Ripa MS, Buse JB. Applying REWIND cardiovascular disease criteria to SUSTAIN 6 and PIONEER 6: An exploratory analysis of cardiovascular outcomes with semaglutide. Diabetes Obes Metab. 2021 Jul;23(7):1677-1680. doi: 10.1111/dom.14360. Epub 2021 Mar 18. PMID 33606902
- [Derived] Husain M, Bain SC, Holst AG, Mark T, Rasmussen S, Lingvay I. Effects of semaglutide on risk of cardiovascular events across a continuum of cardiovascular risk: combined post hoc analysis of the SUSTAIN and PIONEER trials. Cardiovasc Diabetol. 2020 Sep 30;19(1):156. doi: 10.1186/s12933-020-01106-4. PMID 32998732
- [Derived] Thethi TK, Pratley R, Meier JJ. Efficacy, safety and cardiovascular outcomes of once-daily oral semaglutide in patients with type 2 diabetes: The PIONEER programme. Diabetes Obes Metab. 2020 Aug;22(8):1263-1277. doi: 10.1111/dom.14054. Epub 2020 May 13. PMID 32267058
- [Derived] Husain M, Bain SC, Jeppesen OK, Lingvay I, Sorrig R, Treppendahl MB, Vilsboll T. Semaglutide (SUSTAIN and PIONEER) reduces cardiovascular events in type 2 diabetes across varying cardiovascular risk. Diabetes Obes Metab. 2020 Mar;22(3):442-451. doi: 10.1111/dom.13955. Epub 2020 Feb 5. PMID 31903692
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 214 sites in 21 countries: Algeria (4), Argentina (6), Brazil (1), Canada (7), Denmark (5), Germany (10), India (16), Israel (8), Italy (7), Malaysia (10), Mexico (6), Netherlands (5), Poland (5), Romania (8), South Africa (9), Spain (9), Taiwan (4), Thailand (7), Turkey (9) and United Kingdom (9), United Stated (69).
Pre-assignment Details: Data presented in "participant flow" is based on the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Groups:
- Oral Semaglutide: Participants were to take once-daily semaglutide tablets in a dose escalation manner for upto 82 weeks: 3 mg from week 0 to week 4, 7 mg from week 4 to week 8 and 14 mg from week 9 to upto week 82.
- Placebo: Participants were to take oral semaglutide placebo tablets once-daily for a period of upto 82 weeks.
Period: Overall Study
Arm/Group | Oral Semaglutide | Placebo
Started | 1591 | 1592
Full Analysis Set (FAS) | 1591 | 1592
Exposed | 1591 | 1591
Completed | 1586 | 1586
Not Completed | 5 | 6
Not completed — Lost to Follow-up | 2 | 5
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Semaglutide | Placebo | Total
Number analyzed (Participants) | 1591 | 1592 | 3183
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (7) | 66 (7) | 66 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 507 | 500 | 1007
  Male | 1084 | 1092 | 2176
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 253 | 261 | 514
  Not Hispanic or Latino | 1338 | 1331 | 2669
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1148 | 1152 | 2300
  Black or African American | 89 | 103 | 192
  Asian | 324 | 306 | 630
  American Indian or Alaska native | 14 | 15 | 29
  Native Hawaiian or Other Pacific Islander | 5 | 1 | 6
  Other | 11 | 15 | 26
Baseline cardiovasular disease (CVD)/chronic kidney disease (CKD) risk details [Count of Participants; unit: Participants] — This table describes the baseline details of subjects in the study with the risk of CVD and/or CKD.
  Participants
    Established CVD and/or CKD, age ≥ 50 years | 1350 | 1345 | 2695
    Evidence of CV risk factors, age ≥ 60 years | 241 | 247 | 488

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomisation to First Occurrence of a Major Adverse Cardiovascular Event (MACE) Composite Endpoint Consisting of: Cardiovascular Death, Non-fatal Myocardial Infarction or Non-fatal Stroke
Description: Number of participants experiencing a first event of a MACE, defined as cardiovascular death, non-fatal myocardial infarction, or non-fatal stroke are presented. Results are based on the in-trial observation period which started at the date of randomisation, included the period after permanent trial product discontinuation, if any and ended at the date of the follow-up visit regardless of adherence to treatment.
Time Frame: Maximum treatment duration is dependent on event rates and is estimated to be no longer than 19 months + 5 weeks of follow-up period.
Population: Overall number of participants analyzed = full analysis set (FAS) which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 1591 | 1592
Participants | 61 | 76
Statistical Analysis 1: Comparison: Oral Semaglutide vs Placebo; Data from the in-trial observation period. Time from randomisation to first event adjudication committee (EAC) confirmed MACE was analysed using a Cox proportional hazards model with treatment as categorical fixed factor and stratified by evidence of cardiovascular disease at screening. Participants were censored at the end of their in-trial observation period; Test type: Non-Inferiority — This hypothesis was controlled for multiplicity. Non-inferiority of oral semaglutide versus placebo was considered confirmed if the upper limit of the two-sided 95% confidence interval for the HR was strictly below 1.8; p < 0.0001, Regression, Cox — Unadjusted two-sided p-value for test of no difference from the non-inferiority margin (non-inferiority); Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.57 to 1.11]
Statistical Analysis 2: Comparison: Oral Semaglutide vs Placebo; Data from the in-trial observation period. Time from randomisation to first EAC-confirmed MACE was analysed using a Cox proportional hazards model with treatment as categorical fixed factor and stratified by evidence of cardiovascular disease at screening. Participants were censored at the end of their in-trial observation period; Test type: Superiority — This hypothesis was controlled for multiplicity; p = 0.1749, Regression, Cox — Unadjusted two-sided p-value from test of no difference from 1 (superiority); Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.57 to 1.11]

2. Secondary Outcome: Time From Randomisation to First Occurrence of an Expanded Composite Cardiovascular Endpoint Consisting of: Cardiovascular Death, Non-fatal Myocardial Infarction, Non-fatal Stroke, UAP Requiring Hospitalisation or Hospitalisation for Heart Failure
Description: Participants experiencing first occurrence of an expanded composite CV endpoint [defined as cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, UAP (unstable angina pectoris) requiring hospitalisation or heart failure requiring hospitalisation] are presented. Results are based on the in-trial observation period which started at the date of randomisation, included the period after permanent trial product discontinuation, if any and ended at the date of the follow-up visit regardless of adherence to treatment.
Time Frame: as for outcome 1
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 1591 | 1592
Participants | 83 | 100
Statistical Analysis 1: Comparison: Oral Semaglutide vs Placebo; Data from the in-trial observation period. Time from randomisation to first EAC-confirmed expanded cardiovascular outcome was analysed using a Cox proportional hazards model with treatment as categorical fixed factor and stratified by evidence of cardiovascular disease at screening. Participants were censored at the end of their in-trial observation period; Test type: Other — This hypothesis was not controlled for multiplicity; p = 0.1827, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.61 to 1.10]

3. Secondary Outcome: Time From Randomisation to First Occurrence of Each of the Individual Components in the Expanded Composite Cardiovascular Endpoint
Description: Participants experiencing an event onset for each individual component of the expanded composite cardiovascular outcomes (defined as cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, unstable angina requiring hospitalisation or heart failure requiring hospitalisation) are presented. Results are based on the in-trial observation period which started at the date of randomisation, included the period after permanent trial product discontinuation, if any and ended at the date of the follow-up visit regardless of adherence to treatment.
Time Frame: as for outcome 1
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 1591 | 1592
Participants
  Cardiovascular death | 15 | 30
  Non-fatal myocardial infarction | 37 | 31
  Non-fatal stroke | 12 | 16
  Unstable angina requiring hospitalisation | 11 | 7
  Heart failure requiring hospitalisation | 21 | 24
Statistical Analysis 1: Comparison: Oral Semaglutide vs Placebo; Data from the in-trial observation period. Time from randomisation to first EAC-confirmed cardiovascular death (including undetermined cause of death) was analysed using a Cox proportional hazards model with treatment as categorical fixed factor and stratified by evidence of cardiovascular disease at screening. Participants were censored at the end of their in-trial observation period; Test type: Other — This hypothesis was not controlled for multiplicity; p = 0.0261, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.27 to 0.92]
Statistical Analysis 2: Comparison: Oral Semaglutide vs Placebo; Data from the in-trial observation period. Time from randomisation to first EAC-confirmed non-fatal myocardial infarction was analysed using a Cox proportional hazards model with treatment as categorical fixed factor and stratified by evidence of cardiovascular disease at screening. Participants were censored at the end of their in-trial observation period; Test type: Other — This hypothesis was not controlled for multiplicity; p = 0.5044, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.73 to 1.90]
Statistical Analysis 3: Comparison: Oral Semaglutide vs Placebo; Data from the in-trial observation period. Time from randomisation to first EAC-confirmed non-fatal stroke was analysed using a Cox proportional hazards model with treatment as categorical fixed factor and stratified by evidence of cardiovascular disease at screening. Participants were censored at the end of their in-trial observation period; Test type: Other — This hypothesis was not controlled for multiplicity; p = 0.4350, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.35 to 1.57]
Statistical Analysis 4: Comparison: Oral Semaglutide vs Placebo; Data from the in-trial observation period. Time from randomisation to first EAC-confirmed unstable angina pectoris requiring hospitalisation was analysed using a Cox proportional hazards model with treatment as categorical fixed factor and stratified by evidence of cardiovascular disease at screening. Participants were censored at the end of their in-trial observation period; Test type: Other — This hypothesis was not controlled for multiplicity; p = 0.3605, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 1.56, 95% CI 2-sided [0.60 to 4.01]
Statistical Analysis 5: Comparison: Oral Semaglutide vs Placebo; Data from the in-trial observation period. Time from randomisation to first EAC-confirmed hospitalisation for heart failure was analysed using a Cox proportional hazards model with treatment as categorical fixed factor and stratified by evidence of cardiovascular disease at screening. Participants were censored at the end of their in-trial observation period; Test type: Other — This hypothesis was not controlled for multiplicity; p = 0.6227, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.48 to 1.55]

4. Secondary Outcome: Time From Randomisation to First Occurrence of a Composite Endpoint Consisting of: All-cause Death, Non-fatal Myocardial Infarction or Nonfatal Stroke
Description: Participants experiencing first occurrence of a composite CV endpoint (defined as all-cause death, non-fatal myocardial infarction or nonfatal stroke) are presented. Results are based on the in-trial observation period which started at the date of randomisation, included the period after permanent trial product discontinuation, if any and ended at the date of the follow-up visit regardless of adherence to treatment.
Time Frame: as for outcome 1
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 1591 | 1592
Participants | 69 | 89
Statistical Analysis 1: Comparison: Oral Semaglutide vs Placebo; Data from the in-trial observation period. Time from randomisation to first EAC-confirmed all-cause death, non-fatal myocardial infarction or non-fatal stroke was analysed using a Cox proportional hazards model with treatment as categorical fixed factor and stratified by evidence of cardiovascular disease at screening. Participants were censored at the end of their in-trial observation period; Test type: Other — This hypothesis was not controlled for multiplicity; p = 0.0952, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.56 to 1.05]

5. Secondary Outcome: Time From Randomisation to First Occurrence of Fatal or Non-fatal Myocardial Infarction
Description: Number of participants experiencing a first event of a fatal or non-fatal myocardial infarction are presented. Results are based on the in-trial observation period which started at the date of randomisation, included the period after permanent trial product discontinuation, if any and ended at the date of the follow-up visit regardless of adherence to treatment.
Time Frame: as for outcome 1
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 1591 | 1592
Participants | 37 | 35
Statistical Analysis 1: Comparison: Oral Semaglutide vs Placebo; Data from the on-treatment observation period. Time from first dose of trial product to first EAC-confirmed fatal or non-fatal myocardial infarction was analysed using a Cox proportional hazards model with treatment as categorical fixed factor and stratified by evidence of cardiovascular disease at screening. Participants were censored at the end of their on-treatment observation period; Test type: Other — This hypothesis was not controlled for multiplicity; p = 0.8583, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.66 to 1.66]

6. Secondary Outcome: Time From Randomisation to First Occurrence of Fatal or Non-fatal Stroke
Description: Number of participants experiencing a first event of a fatal or non-fatal stroke are presented. Results are based on the in-trial observation period which started at the date of randomisation, included the period after permanent trial product discontinuation, if any and ended at the date of the follow-up visit regardless of adherence to treatment.
Time Frame: as for outcome 1
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 1591 | 1592
Participants | 13 | 17
Statistical Analysis 1: Comparison: Oral Semaglutide vs Placebo; Data from the in-trial observation period. Time from randomisation to first EAC-confirmed fatal or non-fatal stroke was analysed using a Cox proportional hazards model with treatment as categorical fixed factor and stratified by evidence of cardiovascular disease at screening. Participants were censored at the end of their in-trial observation period; Test type: Other — This hypothesis was not controlled for multiplicity; p = 0.4485, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.37 to 1.56]

7. Secondary Outcome: Time From Randomisation to All-cause Death
Description: Number of all-cause deaths in the study are presented. Results are based on the in-trial observation period which started at the date of randomisation, included the period after permanent trial product discontinuation, if any and ended at the date of the follow-up visit regardless of adherence to treatment.
Time Frame: Maximum treatment duration is dependent on event rates and is expected to be no longer than 19 months + 5 weeks of follow-up period.
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 1591 | 1592
Participants | 23 | 45
Statistical Analysis 1: Comparison: Oral Semaglutide vs Placebo; Data from the in-trial observation period. Time from randomisation to first EAC-confirmed all-cause death was analysed using a Cox proportional hazards model with treatment as categorical fixed factor and stratified by evidence of cardiovascular disease at screening. Participants were censored at the end of their in-trial observation period; Test type: Other — This hypothesis was not controlled for multiplicity; p = 0.0078, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.31 to 0.84]

8. Secondary Outcome: Time to First AE Leading to Permanent Trial Product Discontinuation
Description: Number of participants who permanently discontinued trial product in ths study are presented. Results are based on the on-treatment observation period which starts at the date of first dose on trial product; ends on last date on trial product +38 days (ascertainment window).
Time Frame: Maximum treatment duration is dependent on event rates and is expected to be no longer than 19 months + 38 days of ascertainment window.
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 1591 | 1592
Participants | 184 | 104
Statistical Analysis 1: Comparison: Oral Semaglutide vs Placebo; Data from date of first dose of trial product to date of end of treatment visit. Time from first dose to first AE leading to permanent trial product discontinuation was analysed using a Cox proportional hazards model with treatment as categorical fixed factor and stratified by evidence of cardiovascular disease at screening. Participants were censored at the date of their end of treatment visit or at their end of study date, whichever came first; Test type: Other — This hypothesis was not controlled for multiplicity; p < 0.0001, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 1.81, 95% CI 2-sided [1.42 to 2.30]

9. Secondary Outcome: Number of Serious Adverse Events
Description: Number of serious adverse events were recorded from week 0 to week 87 in the study. Results are based on the on-treatment observation period which started at the date of first dose on trial product and ended on last date on trial product +38 days (ascertainment window).
Time Frame: as for outcome 8
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Number; unit: Events
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 1591 | 1592
Events | 545 | 618

10. Secondary Outcome: Change in Eye Examination Category
Description: Participants with eye examination findings, normal, abnormal non clinically significant (NCS) and abnormal clinically significant (CS) at baseline (week -3) and end of treatment visit (week 83) are presented. Results are based on the in-trial observation period which started at the date of randomisation, included the period after permanent trial product discontinuation, if any and ended at the date of the follow-up visit regardless of adherence to treatment.
Time Frame: Week -3, End of treatment
Population: Overall number of participants analyzed = FAS which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 1591 | 1592
Participants
  Left eye fundoscopy (week -3): Normal: number analyzed (Participants) | 1591 | 1590
  Left eye fundoscopy (week -3): Normal | 848 | 843
  Left eye fundoscopy (week -3): Abnormal NCS: number analyzed (Participants) | 1591 | 1590
  Left eye fundoscopy (week -3): Abnormal NCS | 657 | 673
  Left eye fundoscopy (week -3): Abnormal CS: number analyzed (Participants) | 1591 | 1590
  Left eye fundoscopy (week -3): Abnormal CS | 86 | 74
  Right eye fundoscopy (week -3): Normal: number analyzed (Participants) | 1590 | 1591
  Right eye fundoscopy (week -3): Normal | 845 | 858
  Right eye fundoscopy (week -3): Abnormal NCS: number analyzed (Participants) | 1590 | 1591
  Right eye fundoscopy (week -3): Abnormal NCS | 659 | 661
  Right eye fundoscopy (week -3): Abnormal CS: number analyzed (Participants) | 1590 | 1591
  Right eye fundoscopy (week -3): Abnormal CS | 86 | 72
  Left eye fundoscopy (EOT): Normal: number analyzed (Participants) | 1465 | 1449
  Left eye fundoscopy (EOT): Normal | 783 | 790
  Left eye fundoscopy (EOT): Abnormal NCS: number analyzed (Participants) | 1465 | 1449
  Left eye fundoscopy (EOT): Abnormal NCS | 599 | 597
  Left eye fundoscopy (EOT): Abnormal CS: number analyzed (Participants) | 1465 | 1449
  Left eye fundoscopy (EOT): Abnormal CS | 83 | 62
  Right eye fundoscopy (EOT): Normal: number analyzed (Participants) | 1462 | 1450
  Right eye fundoscopy (EOT): Normal | 780 | 787
  Right eye fundoscopy (EOT): Abnormal NCS: number analyzed (Participants) | 1462 | 1450
  Right eye fundoscopy (EOT): Abnormal NCS | 601 | 599
  Right eye fundoscopy (EOT): Abnormal CS: number analyzed (Participants) | 1462 | 1450
  Right eye fundoscopy (EOT): Abnormal CS | 81 | 64

11. Secondary Outcome: Change in Pulse Rate
Description: Change from baseline (week 0) in pulse rate measured at the end of treatment visit (week 83) is reported. Results are based on the on-treatment observation period which started at the date of first dose on trial product, ended on last date on trial product +38 days (ascertainment window).
Time Frame: Week 0, End of treatment
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 1345 | 1411
Beats/minute | 4 (11) | -0 (11)

12. Secondary Outcome: Change in Systolic and Diastolic Blood Pressure
Description: Change from baseline (week 0) in systolic and diastolic blood pressure measured at the end of treatment visit (week 83) is reported. Results are based on the on-treatment observation period which started at the date of first dose on trial product, ended on last date on trial product +38 days (ascertainment window).
Time Frame: Week 0, End of treatment
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 1345 | 1411
mmHg
  Systolic blood pressure | -5 (18) | -2 (18)
  Diastolic blood pressure | -1 (11) | -2 (10)

13. Secondary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline (week 0) in HbA1c measured at the end of treatment visit (week 83) is reported. Results are based on the in-trial observation period which started at the date of randomisation, included the period after permanent trial product discontinuation, if any and ended at the date of the follow-up visit regardless of adherence to treatment.
Time Frame: Week 0, End of treatment
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 1489 | 1473
Percentage of HbA1c | -1.0 (1.4) | -0.3 (1.3)

14. Secondary Outcome: Change in Body Weight
Description: Change from baseline (week 0) in body weight measured at the end of treatment visit (week 83) is reported. Results are based on the in-trial observation period which started at the date of randomisation, included the period after permanent trial product discontinuation, if any and ended at the date of the follow-up visit regardless of adherence to treatment.
Time Frame: Week 0, End of treatment
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 1510 | 1493
Kg | -4.2 (5.7) | -0.8 (4.5)

15. Secondary Outcome: Change in Total Cholesterol - Ratio to Baseline
Description: Change from baseline (week 0) in total cholesterol (mmol/L) at the end of treatment (week 83) visit is presented as ratio to baseline. Results are based on the in-trial observation period which started at the date of randomisation, included the period after permanent trial product discontinuation, if any and ended at the date of the follow-up visit regardless of adherence to treatment.
Time Frame: Week 0, End of treatment
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 1472 | 1469
Ratio of total cholesterol | 0.97 (21.9) | 0.98 (21.1)

16. Secondary Outcome: Change in LDL-cholesterol - Ratio to Baseline
Description: Change from baseline (week 0) in LDL cholesterol (mmol/L) at end of treatment visit (week 83) is presented as ratio to baseline. Results are based on the in-trial observation period which started at the date of randomisation, included the period after permanent trial product discontinuation, if any and ended at the date of the follow-up visit regardless of adherence to treatment.
Time Frame: Week 0, End of treatment
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL-cholesterol
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 1466 | 1467
Ratio of LDL-cholesterol | 0.96 (36.6) | 0.97 (34.5)

17. Secondary Outcome: Change in HDL-cholesterol - Ratio to Baseline
Description: Change from baseline (week 0) in HDL cholesterol (mmol/L) at end of treatment visit (week 83) is presented as ratio to baseline. Results are based on the in-trial observation period which started at the date of randomisation, included the period after permanent trial product discontinuation, if any and ended at the date of the follow-up visit regardless of adherence to treatment.
Time Frame: Week 0, End of treatment
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL-cholesterol
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 1468 | 1467
Ratio of HDL-cholesterol | 1.05 (16.9) | 1.02 (15.9)

18. Secondary Outcome: Change in Triglycerides - Ratio to Baseline
Description: Change from baseline (week 0) in triglycerides (mmol/L) at end of treatment visit (week 83) is presented as ratio to baseline. Results are based on the in-trial observation period which started at the date of randomisation, included the period after permanent trial product discontinuation, if any and ended at the date of the follow-up visit regardless of adherence to treatment.
Time Frame: Week 0, End of treatment
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Oral Semaglutide | Placebo
Number analyzed (Participants) | 1468 | 1467
Ratio of triglycerides | 0.92 (41.8) | 0.97 (39.8)

ADVERSE EVENTS:
Time Frame: Week 0 to 87. SAEs and other AEs were based on the on-treatment observation period, i.e., the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication. All-cause mortality were based on the in-trial observation period, i.e., the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Description: Systematic collection of AEs was limited to SAEs, AEs leading to permanent discontinuation of trial product, medication errors leading to SAEs, severe hypoglycaemic episodes, hepatic events, pregnancies and AEs related to technical complaints and were summarised. Non-serious AEs not fulfilling the above criteria were not systematically collected.
Arm/Group | Oral Semaglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 23/1591 | 45/1591
Serious Adverse Events (participants affected / at risk) | 301/1591 | 358/1591
Other Adverse Events (participants affected / at risk) | 0/1591 | 0/1591
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide (N=1591) | Placebo (N=1591)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 13 (14) | 14 (18)
Acute left ventricular failure (Cardiac disorders) | 2 (2) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 21 (25) | 22 (25)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 8 (9) | 7 (7)
Angina unstable (Cardiac disorders) | 19 (20) | 15 (18)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic aneurysm repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 3 (3) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 6 (8) | 14 (14)
Atrial flutter (Cardiac disorders) | 3 (3) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 3 (3) | 1 (1)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary fistula (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 3 (4)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0)
Carcinoid tumour of the appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 5 (6) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 7 (8)
Cardiac failure acute (Cardiac disorders) | 2 (3) | 2 (2)
Cardiac failure chronic (Cardiac disorders) | 5 (5) | 8 (9)
Cardiac failure congestive (Cardiac disorders) | 9 (12) | 9 (11)
Cardiac flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 3 (3)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 2 (2) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 4 (4) | 4 (5)
Cataract (Eye disorders) | 8 (8) | 5 (6)
Cataract operation (Surgical and medical procedures) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 9 (9) | 7 (7)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 2 (2)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3) | 2 (2)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 4 (4)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 5 (5)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 4 (4)
Clostridium test positive (Investigations) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 9 (9) | 13 (13)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 3 (3)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 1 (1)
Degenerative aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Dementia with Lewy bodies (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 2 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (7)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Drowning (General disorders) | 0 (0) | 1 (1)
Drug dependence (Psychiatric disorders) | 1 (1) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Dyspraxia (Nervous system disorders) | 0 (0) | 1 (1)
Ear injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 3 (3)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 11 (11)
Fatigue (General disorders) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Finger repair operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body in ear (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gallbladder empyema (Infections and infestations) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastric bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (5) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (2)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glaucoma surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Graft haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 2 (3) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Hernia pain (General disorders) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Hypoglycaemic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 9 (11) | 6 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 5 (5) | 3 (3)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
IgA nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Infective tenosynovitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Injection site abscess (Infections and infestations) | 1 (1) | 0 (0)
Injury corneal (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 9 (9) | 11 (12)
Joint arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Lacunar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Latent autoimmune diabetes in adults (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 4 (4)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Light chain disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Ludwig angina (Infections and infestations) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Lumbosacral plexopathy (Nervous system disorders) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Murine typhus (Infections and infestations) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1)
Myelitis (Infections and infestations) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 11 (11) | 9 (9)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 3 (3)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 2 (2)
Neuritis (Nervous system disorders) | 1 (2) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 9 (11) | 7 (9)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Open globe injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 10 (10)
Osteomyelitis (Infections and infestations) | 5 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Pancreatic neuroendocrine tumour metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 7 (7)
Peripheral artery dissection (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 3 (3) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 3 (3)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 3 (3) | 2 (2)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Pneumonia (Infections and infestations) | 12 (13) | 21 (21)
Pneumonia acinetobacter (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia escherichia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural haematuria (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Post procedural pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 2 (2)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Retinopathy proliferative (Eye disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 3 (3) | 6 (6)
Septic shock (Infections and infestations) | 2 (2) | 3 (3)
Sialoadenitis (Infections and infestations) | 0 (0) | 2 (2)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Spinal fusion surgery (Surgical and medical procedures) | 0 (0) | 2 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Splenic haemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Subdural haematoma evacuation (Surgical and medical procedures) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 7 (7) | 4 (4)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 6 (6)
Transurethral prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Trapeziectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 3 (3) | 2 (2)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 5 (5)
Urosepsis (Infections and infestations) | 2 (2) | 3 (5)
VIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Vascular dementia (Nervous system disorders) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Vascular stent restenosis (General disorders) | 0 (0) | 1 (1)
Vasculitic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Wound sepsis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/16/NCT02692716/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/16/NCT02692716/SAP_001.pdf